CLINICAL TRIAL: NCT05052034
Title: Musical Flow for Decreasing Dental Anxiety During Oral and Implants Surgery in COVID-19: a Randomized Controlled Study
Brief Title: Music for Decreasing Dental Anxiety During Oral Surgery in Coronavirus Disease 2019 (COVID-19)
Status: Completed | Type: Observational
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Lorenzo Ángel Esteban Pellicer, Esteban LA, European University of Madrid
Other Study IDs: EuropeanUM
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Dental Anxiety; Covid19
Keywords: Oral Implants; Oral Surgery; Dental Anxiety; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BAROQUE MUSIC: This group would listen to baroque music to control their anxiety level during their oral surgeries.
  Interventions: Other: Music
- CLASSICISM MUSIC: this group would listen to classical music to control their anxiety level during their oral surgeries.
  Interventions: Other: Music
- CONTROL GROUP: This group would not listen to music during their oral intervention, acting as a control group.

INTERVENTIONS:
Other: Music — Through headphones, the patients would listen to different types of music during the intervention.
  Groups: BAROQUE MUSIC; CLASSICISM MUSIC

SUMMARY:
Approximately 100 patients undergoing oral surgery will be divided in 3 groups of musical audition to control anxiety: baroque (N=35), classicism (N=35) and control group (N=30). Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate and Oxygen Saturation will be recorded.

DETAILED DESCRIPTION:
The trend towards greater humanization in all fields of medicine encourages the implementation of non-pharmacological therapies in the management and control of pain and anxiety in patients during dental treatments. Some studies estimate this level of anxiety in up to 51% of patients, who would prefer to undergo some type of sedation during dental treatment. This fear or anxiety may have increased during the COVID-19 pandemic.

Scientific evidence recommends the use of music in daily practice to reduce anxiety and even pain. There are several studies comparing different musical styles. Some of them use a song from the so-called "classical music", but none have analyzed the possible benefits between the different stages of this type of music, which spans several centuries of history.

The purpose of this study is to verify the effect of the use of Baroque and Classical music as non-pharmacological therapy on the control of the level of intraoperative anxiety and pain experienced by patients during the COVID-19 pandemic, subjected to dental extractions. and implant placement.

This randomized controlled study would be carried out on approximately 100 patients who need tooth extractions and dental implant placement in private practice. The patients would be divided into 3 groups: baroque music, classicism music and control group. The patients would be correctly informed and would sign their consent to be part of the study. The music would be played through wireless headphones placed on the patient and connected to their respective music list according to the group to be studied. The parameters recorded during four different moments of surgery would be: systolic blood pressure, diastolic blood pressure, heart rate and oxygen saturation. After the treatment, the patient will complete a visual analog scale (VAS) on their level of pain and anxiety experienced before and after the treatment. For all of them, this surgery would be the first performed by the sole operator of the study, to reduce other subjective criteria associated with the level of pain or anxiety. Another operator would collect the data obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Spanish-speaking patients over 18 years of age who require the placement of a single implant or the extraction of a single tooth.

Exclusion Criteria:

1. Patients with mental illness (dementia)
2. Patients with psychiatric disorders
3. Patients under anxiolytic treatment
4. Patients with visual or motor loss or with any disability that makes it impossible to fill in the forms provided and the visual analog scale (VAS).
5. Patients under medical treatment that could interfere with the anesthesia used in oral surgery.
6. All implant surgeries were ruled out in patients requiring any type of bone regeneration, due to their greater morbidity.
7. All oral surgeries requiring a flap, due to their greater morbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients without diseases that limit the performance of surgery, and that require the extraction of a tooth or the placement of a dental implant.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SPB) | SPB was recorded four times during intervention: "before starting the surgery once sitting in the chair", "immediately after anesthetizing", "immediately after introducing the first surgery drill", "immediately before getting up".
  SPB was recorded in mmHg
Diastolic Blood Pressure (DBP) | SPB was recorded four times during intervention: "before starting the surgery once sitting in the chair", "immediately after anesthetizing", "immediately after introducing the first surgery drill", "immediately before getting up".
  DBP was recorded in mmHg
Heart Rate (HR) | HR was recorded four times during intervention: "before starting the surgery once sitting in the chair", "immediately after anesthetizing", "immediately after introducing the first surgery drill", "immediately before getting up".
  HR was recorded in bpm (beats per minute)
Oxygen Saturation (Sp02) | Sp02 was recorded four times during intervention: "before starting the surgery once sitting in the chair", "immediately after anesthetizing", "immediately after introducing the first surgery drill", "immediately before getting up".
  Sp02 was recorded in % (0-100)

SECONDARY OUTCOMES:
Change from Baseline in Anxiety on the 11-point Visual Analog Scale (VAS) | Baseline before starting surgery to the end of surgery approximately 40 minutes later.
  The VAS is a validated instrument to identify anxiety. Possible scores range from 0 (no anxiety) to 10 (worst anxiety possible).
Change from Baseline in Pain on the 11-point Visual Analog Scale (VAS) | Baseline before starting surgery to the end of surgery approximately 40 minutes later.
  The VAS is a validated instrument to identify pain. Possible scores range from 0 (no pain) to 10 (worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Lorenzo, Principal Investigator — European University of Madrid
Locations (1):
- European University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
All of the individual participant data collected during the study could be available since 3 years after publication for anyone who wishes to access the data, signing a data access agreement.